CLINICAL TRIAL: NCT02466217
Title: Clinical and Multi-omics Cross-phenotyping of Patients With Autoimmune and Auto-inflammatory Diseases
Brief Title: Phenomics in Autoimmune and Inflammatory Diseases
Acronym: TRANSIMMUNOM
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Other Study IDs: P141006; 2015-A00558-41 (Other: EUDRACT)
Record Dates: First submitted 2015-05-12; First posted 2015-06-09 (Estimated); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Healthy Volunteer; Rheumatoid Arthritis; Ankylosing Spondylitis; Systemic Lupus Erythematosus/Antiphospholipid Syndrome; FMF; Cryopyrin-Associated Periodic Syndromes /TNF-receptor Associated Periodic Syndrome; Vasculitis; Uveitis; Myositis; Crohn's Disease; Ulcerative Rectocolitis; Type 1 Diabetes; Unclassified IAD Knee and/or Hip Arthritis, Muscular Dystrophy
Keywords: Auto-immune disease; Auto-inflammatory disease; Omics; System biology
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Lupus Erythematosus, Systemic; Antiphospholipid Syndrome; Vasculitis; Uveitis; Myositis; Crohn Disease; Proctocolitis; Diabetes Mellitus, Type 1; Muscular Dystrophies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: AID groups: Rheumatoid Arthritis, Ankylosing Spondylitis, Systemic Lupus Erythematosus/Antiphospholipid Syndrome, FMF, Cryopyrin-Associated Periodic Syndromes (CAPS)/TNF-receptor Associated Periodic Syndrome (TRAPS), Vasculitis, Uveitis, Myositis, Crohn's Disease, Ulcerative colitis, Type 1 Diabetes
  Interventions: Other: 1: AID groups
- 2: Control groups: knee arthritis, hip arthritis, muscular dystrophy, healthy subject
  Interventions: Other: 2: Control groups

INTERVENTIONS:
Other: 1: AID groups — Clinical and Biological investigations
  Groups: 1: AID groups
Other: 2: Control groups — Clinical and Biological investigations
  Groups: 2: Control groups

SUMMARY:
The family of inflammatory/autoimmune systemic diseases (IAD) form a continuum from pure inflammatory diseases to pure autoimmune diseases, encompassing a large panel of inflammatory diseases with some autoimmune components, and vice versa. Cross phenotyping of patients with IAD should be heuristic and help revise the nosography and the understanding of these diseases.

DETAILED DESCRIPTION:
The family of inflammatory/autoimmune systemic diseases (IAD) represents a large group of human diseases. For most if not all of these IAD, the pathophysiological processes or exact causes remain poorly understood. Progresses in molecular understanding of these IAD have led to realize that these are not two distinct categories of diseases. Rather they form a continuum from pure inflammatory diseases to pure autoimmune diseases, encompassing a large panel of inflammatory diseases with some autoimmune components, and vice versa.

Using systems biology, the investigator aims to improve the understanding of these diseases, to identify novel genes/pathways involved, specific or across the diseases, and to discover biomarkers and potential therapeutic targets.

The investigator will study adult patients with at least one of the following IAD: Rheumatoid Arthritis, Ankylosing Spondylitis, Systemic Lupus Erythematosus/Antiphospholipid Syndrome, Familial Mediterranean Fever (FMF), Cryopyrin-Associated Periodic Syndromes (CAPS) /Tumor Necrosis Factor-receptor Associated Periodic Syndrome (TRAPS), Vasculitis, Uveitis, Myositis, Crohn's Disease, Ulcerative colitis, Type 1 Diabetes. This panel will be completed by controls groups: healthy volunteers, and patients with arthritis (knee and/or hip) or muscular dystrophy.

The biological investigations will notably comprise: immunomics (comprehensive evaluation of peripheral blood cell subsets and serum immunoproteomics, including autoantibodies); transcriptomics; Human Leukocyte Antigen (HLA)-phenotyping; genomics; T-Cell Receptor (TCR) sequencing and microbiota studies.

After signing the informed consent, the subject attends only one visit (Day 0) during which all biological samples will be taken and all clinical information collected.

ELIGIBILITY:
Inclusion Criteria:

* Presenting either:

  * one IAD from our list (Rheumatoid Arthritis, Ankylosing Spondylitis, Systemic Lupus Erythematosus/Antiphospholipid Syndrome, FMF, Cryopyrin-Associated Periodic Syndromes (CAPS)/Tumor Necrosis Factor (TNF)-receptor Associated Periodic Syndrome, Vasculitis, Uveitis, Myositis, Crohn's Disease, Ulcerative colitis, Type 1 Diabetes)
  * or an unclassified IAD : a knee and/or hip arthritis or a muscular dystrophy
  * or healthy subject
* Good veins
* Affiliation to a social security system
* Informed consent form, signed by the participant and the investigator, prior all needed examination

Exclusion Criteria:

* For IADs patients

  * Unauthorized treatment (anticancer chemotherapy)
* For Healthy volunteers

  * Contra-indications for donating blood except from age
  * Known history of IAD (eg: Psoriasis)
* Common exclusion criteria:

  * Pregnant woman
  * Still under the exclusion period from another biomedical study
  * Psychiatric or addiction pathology who could interfere with the ability to fulfill the protocol needs or to provide an informed consent
  * Patient under a legal protection
  * Chronic lifelong viral infection unrelated to the pathology
  * Mild infection within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigator will study adult patients with at least one of the following IAD: Rheumatoid Arthritis, Ankylosing Spondylitis, Systemic Lupus Erythematosus/Antiphospholipid Syndrome, FMF, Cryopyrin-Associated Periodic Syndromes (CAPS)/TNF-receptor Associated Periodic Syndrome (TRAPS), Vasculitis, Uveitis, Myositis, Crohn's Disease, Ulcerative colitis, Type 1 Diabetes. This panel will be completed by controls groups: healthy volunteers, and patients with arthritis (knee and/or hip) or muscular dystrophy
Sampling Method: Non-Probability Sample
Enrollment: 537 (Actual)
Dates: Start 2015-07-29 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Total peripheral blood gene expression between patients, expressed as fluorescence intensity | at day 0, no follow-up
  Identification of novel molecular and cellular pathways involved either in specific diseases or across the IAD continuum through a multiparametric approach
Tregs and Tconvs T cell receptor repertoire, expressed as the % of unique TCR sequences | at day 0, no follow-up
  Identification of novel molecular and cellular pathways involved either in specific diseases or across the IAD continuum through a multiparametric approach
HLA type and SNPs expressed as the occurrence events across patients | at day 0, no follow-up
  Identification of novel molecular and cellular pathways involved either in specific diseases or across the IAD continuum through a multiparametric approach
Microbiote species identification expressed as the % of species per family and genus | at day 0, no follow-up
  Identification of novel molecular and cellular pathways involved either in specific diseases or across the IAD continuum through a multiparametric approach
Cytokines and chemokines expressed as fluorescence intensity | at day 0, no follow-up
  Identification of novel molecular and cellular pathways involved either in specific diseases or across the IAD continuum through a multiparametric approach
Immune cells phenotyping expressed as the each cell type % within total PBMCs | at day 0, no follow-up
  Identification of novel molecular and cellular pathways involved either in specific diseases or across the IAD continuum through a multiparametric approach

SECONDARY OUTCOMES:
Changes in gene expression intensity between patients and healthy controls - for each Disease cohorts | at day 0, no follow-up
  Identification of new biomarkers and potential therapeutic by multiscale analysis
Changes in Tregs and Tconvs TCR sequence frequencies between patients and healthy controls - for each Disease cohorts | at day 0, no follow-up
  Identification of new biomarkers and potential therapeutic by multiscale analysis
Characterization of HLA and SNP profiles in patients and healthy controls - for each Disease cohorts | at day 0, no follow-up
  Identification of new biomarkers and potential therapeutic by multiscale analysis
Changes in Microbiote composition between patients and healthy controls - for each Disease cohorts | at day 0, no follow-up
  Identification of new biomarkers and potential therapeutic by multiscale analysis
Changes in cytokines and chemokines expression levels between patients and healthy controls - for each Disease cohorts | at day 0, no follow-up
  Identification of new biomarkers and potential therapeutic by multiscale analysis
Changes in immune cells frequencies between patients and healthy controls - for each Disease cohorts | at day 0, no follow-up
  Identification of new biomarkers and potential therapeutic by multiscale analysis
Identification of specific and common gene expression levels between patients - between Disease cohorts | at day 0, no follow-up
  Identification of new biomarkers and potential therapeutic by multiscale analysis
Identification of specific and common Tregs and Tconvs TCR sequence frequencies between patients - between Disease cohorts | at day 0, no follow-up
  Identification of new biomarkers and potential therapeutic by multiscale analysis
Characterization of specific and common HLA and SNP profiles in patients - between Disease cohorts | at day 0, no follow-up
  Identification of new biomarkers and potential therapeutic by multiscale analysis
Identification of specific and common microbiote composition between patients - between Disease cohorts | at day 0, no follow-up
  Identification of new biomarkers and potential therapeutic by multiscale analysis
Identification of specific and common cytokines and chemokines expression levels between patients - between Disease cohorts | at day 0, no follow-up
  Identification of new biomarkers and potential therapeutic by multiscale analysis
Characterization specific and common variations in immune cells frequencies between patients - between Disease cohorts | at day 0, no follow-up
  Identification of new biomarkers and potential therapeutic by multiscale analysis

CONTACTS AND LOCATIONS:
Overall Officials: David KLATZMANN, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Rhumatologie - Hôpital Saint-Antoine, Paris
  - CIC Paris-Est, Hôpital PITIE SALPETRIERE, Paris

REFERENCES:
- [Derived] Tchitchek N, Binvignat M, Roux A, Pitoiset F, Dubois J, Marguerit G, Saadoun D, Cacoub P, Sellam J, Berenbaum F, Hartemann A, Amouyal C, Lorenzon R, Mariotti-Ferrandiz E, Rosenzwajg M, Klatzmann D. Deep immunophenotyping reveals that autoimmune and autoinflammatory disorders are spread along two immunological axes capturing disease inflammation levels and types. Ann Rheum Dis. 2024 Apr 11;83(5):638-650. doi: 10.1136/ard-2023-225179. PMID 38182406
- [Derived] Lorenzon R, Mariotti-Ferrandiz E, Aheng C, Ribet C, Toumi F, Pitoiset F, Chaara W, Derian N, Johanet C, Drakos I, Harris S, Amselem S, Berenbaum F, Benveniste O, Bodaghi B, Cacoub P, Grateau G, Amouyal C, Hartemann A, Saadoun D, Sellam J, Seksik P, Sokol H, Salem JE, Vicaut E, Six A, Rosenzwajg M, Bernard C, Klatzmann D. Clinical and multi-omics cross-phenotyping of patients with autoimmune and autoinflammatory diseases: the observational TRANSIMMUNOM protocol. BMJ Open. 2018 Aug 30;8(8):e021037. doi: 10.1136/bmjopen-2017-021037. PMID 30166293